CLINICAL TRIAL: NCT01733043
Title: Dexmedetomidine for Sedation in Individuals With Obstructive Sleep Apnea
Brief Title: Sedative Effects in Obstructive Sleep Apnea
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Failure to secure funding
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00033021
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine infusion (Experimental): Dexmedetomidine 0.5 mcg/kg loading dose administered over 20 minutes, followed by 0.6 mcg/kg/hr infusion for 1 hour and 40 minutes
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Normal saline infusions will be administered over 4 hours at rates mimicking the DEX infusion rate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Precedex
  Arms: Dexmedetomidine infusion
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to determine the effect of dexmedetomidine infusion on the Apnea / Hypopnea Index (AHI) of individuals with previously documented obstructive sleep apnea. We hypothesize that dexmedetomidine infusion may reduce the AHI in patients with obstructive sleep apnea (OSA).

ELIGIBILITY:
Inclusion Criteria:

* All individuals who have previously undergone diagnostic polysomnography in the Sleep Lab which documented significant OSA, and who have not undergone any changes that are likely to alter the severity of their condition since the time of their diagnostic sleep study (loss of weight; surgical therapy for OSA; removal of tonsils; discontinuation of medications likely to affect arousal or respiratory function, etc.) are eligible to participate. Subjects will be identified as they complete outpatient sleep studies or from records of previous sleep studies performed in the Duke Sleep Laboratory. After obtaining informed consent, subjects will be screened by history and physical examination, 12-lead electrocardiogram, and comprehensive metabolic profile.

Exclusion Criteria:

* Exclusion criteria will include a history of illicit drug or alcohol dependence, impaired hepatic (aspartate aminotransferase or alanine aminotransferase > 2x upper limit of normal range) or renal function (receiving dialysis or serum creatinine > 1.5 mg/dL), high-grade (> 1st degree) heart block, or known allergy to dexmedetomidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | 8 hour sleep study
  The primary outcome is frequency of apnea or hypopnea as measured by the apnea hypopnea index

SECONDARY OUTCOMES:
Sleep Architecture | During 8 hour sleep study
  Additional measures of sleep architecture will be made: sleep onset latency, duration of time spent in rapid eye movement (REM) and non-rapid eye movement (NREM) sleep, sleep efficiency, and number of arousals

CONTACTS AND LOCATIONS:
Overall Officials: Brian Colin, MD, Principal Investigator — Duke University